CLINICAL TRIAL: NCT03891628
Title: Modified Attachment and Biobehavioral Catch-Up for Mothers and Their Infants
Brief Title: Modified ABC: A Home-based Parenting Program for Opioid-dependent Mothers and Their Infants
Acronym: mABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Mary Dozier, Amy E. du Pont Chair of Child Development, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PSYC412125
Record Dates: First submitted 2019-02-21; First posted 2019-03-27 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Opioid-Related Disorders; Parent-Child Relations; Infant Development; Parenting
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified ABC (Experimental): Modified Attachment and Biobehavioral Catch-Up (14 session in-home intervention with parents and infants present) and Safe Environment for Every Kid (1 to 2 in-home resource visits)
  Interventions: Behavioral: Modified Attachment and Biobehavioral Catch-up
- Modified DEF (Active Comparator): Modified Developmental Education for Families (14 session in-home intervention with parents and infants present) and Safe Environment for Every Kid (1 to 2 in-home resource visits)
  Interventions: Behavioral: Modified Developmental Education for Families

INTERVENTIONS:
Behavioral: Modified Attachment and Biobehavioral Catch-up — Intervention targets include enhancing nurturance and following the child's lead, as well as supporting use of kangaroo care, swaddling, and breastfeeding.
  Other Names: mABC
  Arms: Modified ABC
Behavioral: Modified Developmental Education for Families — Intervention targets include supporting developmental monitoring and parental engagement in activities that promote cognitive and motor development.
  Other Names: mDEF
  Arms: Modified DEF

SUMMARY:
This study will assess the efficacy of the modified Attachment and Biobehavioral Catch-Up Intervention, adapted for use with peripartum mothers receiving medication-assisted treatment for opioid use disorder. The investigators expect that mothers who receive the modified Attachment and Biobehavioral Catch-up Intervention will show more nurturing and sensitive parenting and more adaptive physiological regulation than parents who receive a control intervention. The investigators expect that infants whose mothers receive the modified Attachment and Biobehavioral Catch-up will show better outcomes in attachment, behavior, and physiological regulation compared to infants of parents who receive the control intervention.

DETAILED DESCRIPTION:
Peripartum mothers will be randomly assigned to receive the modified ABC intervention or the control intervention (modified DEF). Hypotheses relate to parent and child outcomes associated with the intervention.

Hypothesis 1: Compared to mothers who receive the control intervention, mothers who receive the ABC intervention will show more nurturing and sensitive parenting, enhanced neural activity during parenting-relevant tasks, and more normative patterns of DNA methylation, autonomic nervous system activity, and cortisol production.

Hypothesis 2: Compared to infants of mothers who receive the control intervention, infants of mothers who receive the ABC intervention will show more organized and secure attachment patterns, better behavioral regulation during stressors, more advanced social-emotional development, and more normative patterns of DNA methylation, autonomic nervous system activity, and cortisol production.

Hypothesis 3: Enhanced maternal sensitivity will mediate effects of the ABC intervention on improved infant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* In third trimester of pregnancy or up to one month postpartum
* Receiving medication-assisted treatment for opioid use disorder

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Maternal sensitivity | Pre-intervention (third trimester of gestation or up to one month postpartum)
  Maternal sensitivity will be coded observationally from maternal interactions with an infant simulator pre-programmed to coo and then cry. Mothers will be coded for sensitivity, nurturance, intrusiveness, detachment, and positive regard, on 5 point scales from 1-Not at all characteristic to 5-Highly characteristic. Higher scores on sensitivity, nurturance, and positive regard represent more positive parenting, whereas higher scores on nurturance and detachment represent less positive parenting.
Maternal sensitivity | Infant age 3 months
  Maternal sensitivity will be coded observationally from mother-infant play interactions, in which mothers will be given toys and asked to play as they normally would. Mothers will be coded for sensitivity, nurturance, intrusiveness, detachment, and positive regard, on 5 point scales from 1-Not at all characteristic to 5-Highly characteristic. Higher scores on sensitivity, nurturance, and positive regard represent more positive parenting, whereas higher scores on nurturance and detachment represent less positive parenting.
Maternal sensitivity | Infant age 6 months
  Maternal sensitivity will be coded observationally from mother-infant play interactions, in which mothers will be given toys and asked to play as they normally would. Mothers will be coded for sensitivity, nurturance, intrusiveness, detachment, and positive regard, on 5 point scales from 1-Not at all characteristic to 5-Highly characteristic. Higher scores on sensitivity, nurturance, and positive regard represent more positive parenting, whereas higher scores on nurturance and detachment represent less positive parenting.
Maternal sensitivity | Infant age 12 months
  Maternal sensitivity will be coded observationally from mother-infant play interactions, in which mothers will be given toys and asked to play as they normally would. Mothers will be coded for sensitivity, nurturance, intrusiveness, detachment, and positive regard, on 5 point scales from 1-Not at all characteristic to 5-Highly characteristic. Higher scores on sensitivity, nurturance, and positive regard represent more positive parenting, whereas higher scores on nurturance and detachment represent less positive parenting.
Maternal methylation of μ-opioid receptor (OPRM1) gene | Pre-intervention (third trimester of gestation or up to one month postpartum)
  Maternal methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva.
Maternal methylation of μ-opioid receptor (OPRM1) gene | Infant age 3 months
  Maternal methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva.
Maternal methylation of μ-opioid receptor (OPRM1) gene | Infant age 6 months
  Maternal methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva.
Maternal methylation of μ-opioid receptor (OPRM1) gene | Infant age 12 months
  Maternal methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva.
Maternal methylation of oxytocin receptor (OXTR) gene | Pre-intervention (third trimester of gestation or up to one month postpartum)
  Maternal methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva.
Maternal methylation of oxytocin receptor (OXTR) gene | Infant age 3 months
  Maternal methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva.
Maternal methylation of oxytocin receptor (OXTR) gene | Infant age 6 months
  Maternal methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva.
Maternal methylation of oxytocin receptor (OXTR) gene | Infant age 12 months
  Maternal methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva.
Infant methylation of μ-opioid receptor (OPRM1) gene | Infant age 3 months
  Infant methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva.
Infant methylation of μ-opioid receptor (OPRM1) gene | Infant age 6 months
  Infant methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva.
Infant methylation of μ-opioid receptor (OPRM1) gene | Infant age 12 months
  Infant methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva.
Infant methylation of oxytocin receptor (OXTR) gene | Infant age 3 months
  Infant methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva.
Infant methylation of oxytocin receptor (OXTR) gene | Infant age 6 months
  Infant methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva.
Infant methylation of oxytocin receptor (OXTR) gene | Infant age 12 months
  Infant methylation will be assessed using direct bisulfite sequencing of DNA extracted from saliva.
Maternal neural activity (EEG) - Own child-other child task | Pre-intervention (third trimester of gestation or up to one month postpartum)
  Maternal event-related potentials will be assessed using electroencephalogram (EEG) while viewing photos of their own infants, familiar infants, and unfamiliar infants.
Maternal neural activity (EEG) - Own child-other child task | Infant age 12 months
  Maternal event-related potentials will be assessed using electroencephalogram (EEG) while viewing photos of their own infants, familiar infants, and unfamiliar infants.
Maternal neural activity (EEG) - Reward sensitivity task | Pre-intervention (third trimester of gestation or up to one month postpartum)
  Maternal event-related potentials will be assessed using electroencephalogram (EEG) while viewing images from four categories: opioid-related images, baby pictures, positive images, and neutral images.
Maternal neural activity (EEG) - Reward sensitivity task | Infant age 12 months
  Maternal event-related potentials will be assessed using electroencephalogram (EEG) while viewing images from four categories: opioid-related images, baby pictures, positive images, and neutral images.
Maternal neural activity (EEG) - Child emotion task | Pre-intervention (third trimester of gestation or up to one month postpartum)
  Maternal event-related potentials will be assessed using electroencephalogram (EEG) while viewing images of children crying, laughing, and showing neutral expressions.
Maternal neural activity (EEG) - Child emotion task | Infant age 12 months
  Maternal event-related potentials will be assessed using electroencephalogram (EEG) while viewing images of children crying, laughing, and showing neutral expressions.
Maternal parasympathetic nervous system activity | Pre-intervention (third trimester of gestation or up to one month postpartum)
  Maternal parasympathetic nervous system activity will be assessed using respiratory sinus arrhythmia.
Maternal sympathetic nervous system activity | Pre-intervention (third trimester of gestation or up to one month postpartum)
  Maternal sympathetic nervous system activity will be assessed using pre-ejection period.
Maternal parasympathetic nervous system activity | Infant age 3 months
  Maternal parasympathetic nervous system activity will be assessed using respiratory sinus arrhythmia.
Maternal sympathetic nervous system activity | Infant age 3 months
  Maternal sympathetic nervous system activity will be assessed using pre-ejection period.
Maternal parasympathetic nervous system activity | Infant age 6 months
  Maternal parasympathetic nervous system activity will be assessed using respiratory sinus arrhythmia.
Maternal sympathetic nervous system activity | Infant age 6 months
  Maternal sympathetic nervous system activity will be assessed using pre-ejection period.
Maternal parasympathetic nervous system activity | Infant age 12 months
  Maternal parasympathetic nervous system activity will be assessed using respiratory sinus arrhythmia.
Maternal sympathetic nervous system activity | Infant age 12 months
  Maternal sympathetic nervous system activity will be assessed using pre-ejection period.
Infant parasympathetic nervous system activity | Infant age 3 months
  Infant parasympathetic nervous system activity will be assessed using respiratory sinus arrhythmia.
Infant sympathetic nervous system activity | Infant age 3 months
  Infant sympathetic nervous system activity will be assessed using pre-ejection period.
Infant parasympathetic nervous system activity | Infant age 6 months
  Infant parasympathetic nervous system activity will be assessed using respiratory sinus arrhythmia.
Infant sympathetic nervous system activity | Infant age 6 months
  Infant sympathetic nervous system activity will be assessed using pre-ejection period.
Infant parasympathetic nervous system activity | Infant age 12 months
  Infant parasympathetic nervous system activity will be assessed using respiratory sinus arrhythmia.
Infant sympathetic nervous system activity | Infant age 12 months
  Infant sympathetic nervous system activity will be assessed using pre-ejection period.
Maternal diurnal cortisol production | Pre-intervention (third trimester of gestation or up to one month postpartum)
  Maternal diurnal cortisol production will be assessed through salivary cortisol levels collected at wake-time and bed-time.
Maternal diurnal cortisol production | Infant age 12 months
  Maternal diurnal cortisol production will be assessed through salivary cortisol levels collected at wake-time and bed-time.
Infant diurnal cortisol production | Infant age 3 months
  Infant diurnal cortisol production will be assessed through salivary cortisol levels collected at wake-time and bed-time.
Infant diurnal cortisol production | Infant age 6 months
  Infant diurnal cortisol production will be assessed through salivary cortisol levels collected at wake-time and bed-time.
Infant diurnal cortisol production | Infant age 12 months
  Infant diurnal cortisol production will be assessed through salivary cortisol levels collected at wake-time and bed-time.
Infant behavioral regulation - Still Face Paradigm | Infant age 6 months
  Behavioral coding of emotion reactivity and regulation will be conducted from video recordings of the Still Face Paradigm, a mild social stressor.
Infant behavioral regulation - Arm Restraint Task | Infant age 12 months
  Behavioral coding of emotion reactivity and regulation will be conducted from video recordings of the Arm Restraint Task, a mild stressor.
Infant attachment | Infant age 12 months
  Infant attachment will be assessed using the Strange Situation.
Infant cognitive development | Infant age 3 months
  Infant cognitive development will be assessed through maternal report on the Ages and Stages Questionnaire.
Infant motor development | Infant age 3 months
  Infant motor development will be assessed through maternal report on the Ages and Stages Questionnaire.
Infant social-emotional development | Infant age 3 months
  Infant social-emotional development will be assessed through maternal report on the Ages and Stages Questionnaire: Social-Emotional.
Infant cognitive development | Infant age 6 months
  Infant cognitive development will be assessed through maternal report on the Ages and Stages Questionnaire.
Infant motor development | Infant age 6 months
  Infant motor development will be assessed through maternal report on the Ages and Stages Questionnaire.
Infant social-emotional development | Infant age 6 months
  Infant social-emotional development will be assessed through maternal report on the Ages and Stages Questionnaire: Social-Emotional.
Infant cognitive development | Infant age 12 months
  Infant cognitive development will be assessed through maternal report on the Ages and Stages Questionnaire.
Infant motor development | Infant age 12 months
  Infant motor development will be assessed through maternal report on the Ages and Stages Questionnaire.
Infant social-emotional development | Infant age 12 months
  Infant social-emotional development will be assessed through maternal report on the Ages and Stages Questionnaire: Social-Emotional.
Infant social-emotional problems | Infant age 12 months
  Infant social-emotional problems will be assessed through maternal report on the Brief Infant-Toddler Social Emotional Assessment.
Maternal self-efficacy | Pre-intervention (third trimester of gestation or up to one month postpartum)
  Mothers will report on their parenting self-efficacy using the Maternal Self-Efficacy Scale. Mothers will rate their self-efficacy for each of ten items (nine discrete parenting behaviors and one global parenting item) on a 4-point scale from 1-not good at all to 4-very good. Scores are summed to form a total maternal self-efficacy composite (possible range = 10-40), where higher scores indicated more maternal self-efficacy.
Maternal self-efficacy | Infant age 12 months
  Mothers will report on their parenting self-efficacy using the Maternal Self-Efficacy Scale. Mothers will rate their self-efficacy for each of ten items (nine discrete parenting behaviors and one global parenting item) on a 4-point scale from 1-not good at all to 4-very good. Scores are summed to form a total maternal self-efficacy composite (possible range = 10-40), where higher scores indicated more maternal self-efficacy.
Maternal emotion regulation | Pre-intervention (third trimester of gestation or up to one month postpartum)
  Mothers will report on their emotion regulation using the Difficulties with Emotion Regulation Scale - Short Form (DERS-SF). The DERS-SF consists of 18 items rated on a scale from 1-almost never to 5-almost always. The DERS-SF yields six subscales (strategies, non-acceptance, impulse, goals, awareness, and clarity), each of which range from 3 to 15, and one total score, which ranges from 18 to 90. Higher scores indicate greater emotion dysregulation.
Maternal emotion regulation | Infant age 12 months
  Mothers will report on their emotion regulation using the Difficulties with Emotion Regulation Scale - Short Form (DERS-SF). The DERS-SF consists of 18 items rated on a scale from 1-almost never to 5-almost always. The DERS-SF yields six subscales (strategies, non-acceptance, impulse, goals, awareness, and clarity), each of which range from 3 to 15, and one total score, which ranges from 18 to 90. Higher scores indicate greater emotion dysregulation.

SECONDARY OUTCOMES:
Maternal substance use - interview | Pre-intervention (third trimester of gestation or up to one month postpartum)
  The Timeline Followback Interview will be used to assess maternal use of opioids, tobacco, alcohol, marijuana, and other substances.
Maternal substance use - interview | Infant age 6 months
  The Timeline Followback Interview will be used to assess maternal use of opioids, tobacco, alcohol, marijuana, and other substances.
Maternal substance use - interview | Infant age 12 months
  The Timeline Followback Interview will be used to assess maternal use of opioids, tobacco, alcohol, marijuana, and other substances.
Maternal substance use - questionnaire | Pre-intervention (third trimester of gestation or up to one month postpartum)
  Mothers will report their history of substance use using the NIDA ASSIST questionnaire.
Maternal substance use - questionnaire | Infant age 3 months
  Mothers will report recent substance use using the NIDA Quick Screen questionnaire.
Maternal substance use - questionnaire | Infant age 6 months
  Mothers will report recent substance use using the NIDA Quick Screen questionnaire.
Maternal substance use - questionnaire | Infant age 12 months
  Mothers will report recent substance use using the NIDA Quick Screen questionnaire.
Maternal depressive symptoms | Pre-intervention (third trimester of gestation or up to one month postpartum)
  Maternal depressive symptoms will be self-reported using the Beck Depression Inventory.
Maternal depressive symptoms | Infant age 3 months
  Maternal depressive symptoms will be self-reported using the Beck Depression Inventory.
Maternal depressive symptoms | Infant age 6 months
  Maternal depressive symptoms will be self-reported using the Beck Depression Inventory.
Maternal depressive symptoms | Infant age 12 months
  Maternal depressive symptoms will be self-reported using the Beck Depression Inventory.
Infant physical growth | Infant age 3 months
  Infant physical growth will be assessed using weight, length, and head circumference.
Infant physical growth | Infant age 6 months
  Infant physical growth will be assessed using weight, length, and head circumference.
Infant physical growth | Infant age 12 months
  Infant physical growth will be assessed using weight, length, and head circumference.
Maternal experiences during labor and delivery | Infant age 3 months
  Mothers will report on their experiences during labor and delivery using the Birth Satisfaction Scale-Revised questionnaire (BSS-R). This measure consists of ten items rated on a 5-point scale from 1-Strongly Disagree to 5-Strongly Agree. The total score ranges from 10-50, where higher scores represent more birth satisfaction.
Home environment | Infant age 3 months
  The home environment will be assessed using the Cognitive Stimulation subscale of the HOME Short Form, a combination of observation (two items) and maternal report (seven items). Observation items are binary (yes/no), and mother-report items are rated on a Likert-type scale and dichotomized. Dichotomous items are summed to form a total score (range 0-9), with higher scores indicating more cognitive stimulation.
Maternal reward responsiveness | Pre-intervention (third trimester of gestation or up to one month postpartum)
  Mothers will report their reward responsiveness using the Reward Responsiveness Scale. This is an 8-item scale rated on a 4-point scale from 1-Strong Disagreement to 4-Strong Agreement. The total score ranges from 8 to 32, with higher scores representing greater reward responsiveness.
Maternal reward responsiveness | Infant age 12 months
  Mothers will report their reward responsiveness using the Reward Responsiveness Scale. This is an 8-item scale rated on a 4-point scale from 1-Strong Disagreement to 4-Strong Agreement. The total score ranges from 8 to 32, with higher scores representing greater reward responsiveness.
Maternal sleep | Pre-intervention (third trimester of gestation or up to one month postpartum)
  Mothers will report on their sleep habits using the Pittsburgh Sleep Quality Index.
Maternal sleep | Infant age 3 months
  Mothers will report on their sleep habits using the Pittsburgh Sleep Quality Index.
Maternal sleep | Infant age 6 months
  Mothers will report on their sleep habits using the Pittsburgh Sleep Quality Index.
Maternal sleep | Infant age 12 months
  Mothers will report on their sleep habits using the Pittsburgh Sleep Quality Index.
Infant sleep | Infant age 3 months
  Mothers will report on their infant's sleep habits using the Brief Infant Sleep Questionnaire.
Infant sleep | Infant age 6 months
  Mothers will report on their infant's sleep habits using the Brief Infant Sleep Questionnaire.
Infant sleep | Infant age 12 months
  Mothers will report on their infant's sleep habits using the Brief Infant Sleep Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tabachnick AR, Eiden RD, Labella MH, Dozier M. Effects of an attachment-based intervention on autonomic regulation among opioid-exposed infants. Dev Psychobiol. 2022 Sep;64(6):e22286. doi: 10.1002/dev.22286. PMID 35748625